CLINICAL TRIAL: NCT03522870
Title: Effects of Novel Flash Glucose Monitoring System on Glycemic Control in Adult Patients With Type 1 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jianping Weng, Professor,Principal Investigator,Department of Endocrinology and Metabolism，The Third Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017YFC1309601
Record Dates: First submitted 2018-04-18; First posted 2018-05-11 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Flash glucose monitoring system; FGMS
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Flash Glucose Monitoring System (Experimental): People selected to this group will using flash glucose monitoring system continuously on Week 2-14 and Week 14-26.
  Interventions: Device: Flash glucose monitoring system
- SMBG (Active Comparator): People selected to this group will using SMBG continuously on Week 2-14 and Week 14-26.
  Interventions: Device: SMBG

INTERVENTIONS:
Device: Flash glucose monitoring system — Using flash glucose monitoring system continuously on Week 2-14 and Week 14-26
  Other Names: Freestyle Libre®;Abbott Diabetes Care,Witney, Oxon,UK
  Arms: Flash Glucose Monitoring System
Device: SMBG — Performing SMBG at least three times/day on Week 2-14 and Week 14-26
  Other Names: Capillary blood glucose tested by Bayer
  Arms: SMBG

SUMMARY:
This trial is a randomized, multi-center, parallel-group, efficacy and safety study with a 26-weeks follow- up(after 2-week recruitment). The study aims to: 1)compare the effects of novel flash glucose monitoring system (FGMS) and conventional Self Measurement of Blood Glucose (SMBG); and 2) optimize integrated management for glycaemic control in adult patients with type 1 diabetes who are sub-optimally controlled.

DETAILED DESCRIPTION:
Subjects with Type 1 diabetes who meet criteria will be enrolled at up to eight clinical research sites in China. Subjects will be randomized to either flash glucose monitoring system(Freestyle Libre®;Abbott Diabetes Care,Witney, Oxon,UK) or conventional Self Measurement of Blood Glucose (Bayer®)alone at least three times per day. Primary outcome variable is the difference in HbA1c which will be analyzed in a central laboratory between baseline and the 26weeks follow-up. Secondary outcome variables such as time-in-range, frequency and duration of and hyperglycemic episodes etc. will be assessed at baseline (Week 0 to 2), Week 12-14 and Week 24-26 via professional continuous glucose system (Ipro2®; Medtronic). At the same time, demographic factors, clinical data, patient reported outcome (PROs) will be collected. Assessment of Adverse Events will occur via self-reporting at each visit and/or phone call. All patients will receive same ordinary diabetes education.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years and older;
2. Diagnosed with type 1 diabetes with the criteria established by WHO in 1999,with duration more than 1 year;
3. Glycosylated Hemoglobin A1c concentration between 7% and 10%;
4. Self-monitor of blood glucose levels on a regular basis for 2 months previous( at least 3 times per day) and have willing to insist for at least 6 months
5. Using CSII or MDI for at least 3 months, stable diabetes medication regimen for 3 months prior to study entry(change in insulin ≦20%).
6. Willing to wear CGM;
7. Able to speak, read, and write Chinese

Exclusion Criteria:

1. Having used CGM 3 months prior to study entry;
2. Had severe diabetic complications such as PDR in diabetic retinopathy and ESRD of diabetic nephropathy, assessed by investigators;
3. Receiving oral steroid therapy for any disorders and continuous use of paracetamol.
4. Had known allergy to medical-grade adhesives or CGM and its affiliated components;
5. Being pregnant or planning pregnancy (as demonstrated by a positive test at study entry);
6. Recent severe diseases like myocardial infarction,stroke,psychiatric diseases(historical/recent),malignant tumor, kidney disease(defined as eGFR<45), dermatosis, decided by investigator.
7. Current participation in another investigational study (must have completed any previous studies at least 30 days prior to being enrolled in this study);
8. Currently abusing illicit drugs, alcohol, or prescription drugs;
9. Any condition that could impact reliability of the HbA1C measurement,（e.g.hemoglobinopathy, hemolytic anemia, chronic liver disease),decided by investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2022-06-19 (Actual); Study Completion 2022-06-19 (Actual)

PRIMARY OUTCOMES:
Glycosylated Hemoglobin A1c | baseline,week14,week26
  Difference in HbA1c at week 14 and week26 adjusted for baseline(week 0)

SECONDARY OUTCOMES:
Time in Range | baseline,week12-14,week24-26
  Difference in time in Range (70-180 mg/dL) assessed in week 12-14 and week 24-26 adjusted for baseline(week 0 to 2)
Time in Hypoglycemia | baseline,week12-14,week24-26
  Difference in time in hypoglycaemia (<70mg/dL,<54mg/dL and<40mg/dL) assessed in week 12-14 and week 24-26 adjusted for baseline(week 0 to 2)
Time in Hyperglycaemia | baseline,week12-14,week24-26
  Difference in time in hyperglycaemia (>180mg/dL and>300mg/dL) assessed in week 12-14 and week 24-26 adjusted for baseline(week 0 to 2)
Percentage of HbA1c in Range | baseline,week14,week26
  Difference in Percentage of HbA1c at week14 and week 26 adjusted for baseline(week 0)
Standard deviation of glucose | baseline,week12-14,week24-26
  Difference in standard deviation of glucose assessed in week 12-14 and week 24-26 adjusted for baseline(week 0 to 2)
Mean glucose levels | baseline,week12-14,week24-26
  Difference in mean glucose levels assessed in week 12-14 and week 24-26 adjusted for baseline(week0 to 2)
The area under the curve of hypoglycemia/ hyperglycaemia | baseline,week12-14,week24-26
Frequency in hypoglycemia/ hyperglycaemia | baseline,week12-14,week24-26
Frequency in severe hypoglycaemia | baseline,week12-14,week24-26
Frequency in adverse events about device | 26weeks
Frequency in using FGM | 24 weeks
Frequency in SMBG | 26 weeks
Total daily dose of insulin | 26 weeks
The Diabetes Distress Scale (DDS) | baseline,week 14 and week 26
  The Chinese version of the Diabetes Distress Scale is to evaluate diabetes-related emotional distress in Chinses diabetic patients. The scale consists of 17 items, contains four domains including emotional burden sub-scale, physician-related distress subscale, regimen-related distress subscale, and diabetes-related interpersonal distress. Each item is rated on a 6-point Likert scale from 1(no problem) to 6(serious problem). An average score ≥3 is the cut-off point which is considered to more than moderate problem. Administration time is approximately 10 minutes.
Hypoglycaemia Fear Scale(HFS) | baseline,week 14 and week 26
  The Chinses version of Hypoglycemia Fear Survey II- Worry Scale (CHFSII-WS) is to evaluate psychological status for diabetic patients. Change in Hypoglycemia Fear Scale (HFS) score will be assessed in week 14 and week 26 adjusted for baseline(week0). These validated surveys consist of 18 questions which measure dimensions of anxiety and fear surrounding hypoglycemia. Each item is rated on 5-point Likert scale from 0(never related) to 4(very related). "Never relative" scores 1, and so on and so forth, and "very related" scores 4. Patients with higher scores are considered with more anxieties and fear of hypoglycemia. Administration time is approximately 10 minutes.
EQ-5D-5L | baseline,week 14 and week 26
  The Chinese version of the EQ-5D-5L is widely used to evaluate quality of life. The EQ-5D-5L is converted to a single summary index by applying a formula that essentially attaches weights to each of the levels in each dimension. The formula is based on the valuation of EQ-5D health states from general population samples. It contains the health description system and Visual Analogue Score (VAS). The health description system includes 5 dimensions including mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each item is rated on 5 levels from 1(no problems) to 5(extreme problem). And the EQ-VAS is to evaluate the health condition assessed by patients. The top score (100) means the best health conditions and the bottom one (0) means the worst. Administration time is approximately 3minutes. Difference in EQ-5D-5Ls assessed in week 14 and week26 adjusted for baseline(week0-2).

CONTACTS AND LOCATIONS:
Overall Officials: Xueying Zheng, MD, Principal Investigator — The First Affiliated Hospital of USTC; Jing Lu, PHD, Principal Investigator — Department of Endocrinology, Nanjing Drum Tower Hospital Affiliated to Nanjing University Medical School, Nanjing, China.
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Zhou Y, Deng H, Liu H, Yang D, Xu W, Yao B, Yan J, Weng J. Effects of novel flash glucose monitoring system on glycaemic control in adult patients with type 1 diabetes mellitus: protocol of a multicentre randomised controlled trial. BMJ Open. 2020 Dec 4;10(12):e039400. doi: 10.1136/bmjopen-2020-039400. PMID 33277281
- [Result] Liu H, Yang D, Deng H, Xu W, Lv J, Zhou Y, Luo S, Zheng X, Liang H, Yao B, Qiu L, Wang F, Liu F, Yan J, Weng J. Impacts of glycemic variability on the relationship between glucose management indicator from iPro2 and laboratory hemoglobin A1c in adult patients with type 1 diabetes mellitus. Ther Adv Endocrinol Metab. 2020 Jun 8;11:2042018820931664. doi: 10.1177/2042018820931664. eCollection 2020. PMID 32551036
- [Result] Yan J, Zhou Y, Zheng X, Zheng M, Lu J, Luo S, Yang D, Deng H, Xu W, Bi Y, Bao W, Weng J. Effects of intermittently scanned continuous glucose monitoring in adult type 1 diabetes patients with suboptimal glycaemic control: A multi-centre randomized controlled trial. Diabetes Metab Res Rev. 2023 May;39(4):e3614. doi: 10.1002/dmrr.3614. Epub 2023 Feb 7. PMID 36670050
- [Result] Zhou Y, Mai X, Deng H, Yang D, Zheng M, Huang B, Xu L, Weng J, Xu W, Yan J. Discrepancies in glycemic metrics derived from different continuous glucose monitoring systems in adult patients with type 1 diabetes mellitus. J Diabetes. 2022 Jul;14(7):476-484. doi: 10.1111/1753-0407.13296. Epub 2022 Jul 21. PMID 35864804